CLINICAL TRIAL: NCT03085888
Title: The STRIVE Study: Breast Cancer Screening Cohort for the Development of Assays for Early Cancer Detection
Brief Title: The STRIVE Study: Development of a Blood Test for Early Detection of Multiple Cancer Types
Status: Completed | Type: Observational
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GRAIL-002
Record Dates: First submitted 2017-01-17; First posted 2017-03-21 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms; Cancer
Keywords: Cancer Screening; High-Throughput Nucleotide Sequencing; Deep Sequencing; Circulating cell-free tumor DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: This is a prospectively enrolling cohort study with a pre-specified molecular analysis plan. A stratified case-cohort design will be employed to select cancer cases and non-cancer subjects who will be assayed. All cases of cancer (breast and non-breast cancer) will be selected. A random subset of the overall study cohort will also be selected.

SUMMARY:
GRAIL is using high-intensity sequencing of circulating cell-free nucleic acids (cfNAs) to develop blood tests to detect cancer early. The purpose of this study is to validate the ability of the pre-specified GRAIL Test to detect breast cancer and other invasive cancers, including hematologic malignancies, that will occur within one year of the first study blood draw.

DETAILED DESCRIPTION:
Detection of early stage cancer may be possible through analysis of circulating cell-free nucleic acids (cfNAs) shed into the blood by tumors. GRAIL is using high-intensity sequencing (based on broad genomic coverage and deep sequencing) of cfNAs, combined with machine learning, to develop blood tests to detect cancer early. The purpose of this prospective, multi-center, observational cohort study is to validate an assay for the early detection of breast cancer and other invasive cancers, including hematologic malignancies. The study will collect blood samples from participants within 28 days of their screening mammogram. Additional blood samples will also be collected for a subset of participants. For participants who receive a cancer diagnosis during the study, archival tissue samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing mammography for screening indications or have an appointment for screening mammography.
2. Participant provides informed consent and expresses understanding of the protocol and its requirements, risks, and discomforts.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This multi-center study aims to enroll approximately 100,000 women undergoing mammography for screening indications and associated medical care from participating study centers.
Sampling Method: Non-Probability Sample
Enrollment: 99481 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of the pre-specified GRAIL Test to detect invasive cancers (including hematologic malignancies). | From date of first blood draw until first documented invasive cancer diagnosis, assessed up to 30 Months
To refine the predictive algorithms and cut points of the GRAIL test to detect breast and other invasive cancers (including hematologic malignancies). | From date of first blood draw until first documented invasive cancer diagnosis, assessed up to 30 Months

SECONDARY OUTCOMES:
Diagnosis of invasive cancers, including hematologic malignancies, diagnosed in To evaluate the performance of the GRAIL Test to detect invasive cancers in clinically meaningful subgroups. | From date of first blood draw until first documented invasive cancer diagnosis, assessed up to 30 Months
  sequencing to characterize cfNA profiles.
Diagnosis of invasive cancers, including hematologic malignancies, diagnosed in 6-month time windows (e.g. 0-6 months, >6-12 months, >12-18 months, >18-24 months). | From date of first blood draw until first documented invasive cancer diagnosis, assessed up to 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: GRAIL Study Director, Study Director — GRAIL, Inc.
Locations (34):
- United States (34):
  - Mayo Clinic, Phoenix, Arizona
  - Scottsdale Medical Imaging Research, Scottsdale, Arizona
  - Sutter Health, Elk Grove, California
  - Sutter Health, Folsom, California
  - Sutter Health, Mountain View, California
  - Sutter Health, Oakland, California
  - Sutter Health, Palo Alto, California
  - Sutter Health, Roseville, California
  - Sutter Health, Sacramento, California
  - Sutter Health, San Francisco, California
  - Sutter Health, San Mateo, California
  - Sutter Health, Santa Cruz, California
  - Sutter Health, Santa Rosa, California
  - Mayo Clinic, Jacksonville, Florida
  - Sarah Cannon Research Institute, Snellville, Georgia
  - Sarah Cannon Research Institute, Overland Park, Kansas
  - Henry Ford Health System, Dearborn, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Health System, Grosse Pointe Farms, Michigan
  - Henry Ford Health System, Livonia, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Sarah Cannon Research Institute, Independence, Missouri
  - Cleveland Clinic, Avon, Ohio
  - Cleveland Clinic, Beachwood, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Sarah Cannon Research Institute, Charleston, South Carolina
  - Sarah Cannon Research Institute, Hermitage, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Sarah Cannon Research Institute, McKinney, Texas
  - Sarah Cannon Research Institute, Salt Lake City, Utah
  - Sarah Cannon Research Institute, Richmond, Virginia
  - Sarah Cannon Research Institute, Salem, Virginia
  - Mayo Clinic, Eau Claire, Wisconsin
  - Mayo Clinic, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766